CLINICAL TRIAL: NCT03829085
Title: Randomized Multicenter Prospective Clinical Trial to Compare the Effectiveness of Starting Early Oral Diet Versus Nil Per Oral in Patients With Acute Pancreatitis
Brief Title: Study of the Diet in Patients With the Diagnostic of Acute Pancreatitis
Acronym: PADI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Garraf (Other)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Elena Ramírez-Maldonado, Principal investigator, Consorci Sanitari del Garraf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PADI_01
Record Dates: First submitted 2019-01-27; First posted 2019-02-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pancreatitis, Acute
Keywords: Acute Pancreatitis; Oral refeeding; Nutrition; Length hospitalization
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early oral refeeding (Active Comparator): The patients will be started the oral refeeding from the first day of admission in the hospital.
  Patients will receive a low fat solid diet with more and less 1500 calories, 35 g fat day
  Interventions: Other: EARLY ORAL REFEEDING
- FASTING (No Intervention): The oral diet will be reintroduced in a traditional stepwise manner until the symptoms, signs, inflammatory parameters of AP have resolved

INTERVENTIONS:
Other: EARLY ORAL REFEEDING — the oral refeeding will be started after admission. Patients will receive a low fat solid diet with more and less 1500 calories, 35 g fat day
  Arms: Early oral refeeding

SUMMARY:
Acute pancreatitis (AP) is a common condition in emergency services worldwide. Approximately 85% of AP are mild and the patients usually recover within 1 to 2 weeks, not requeiring any critical care and organ support. The management of mild AP conventionally involves fasting, intravenous hydration and adequate analgesia until pain improves in order to prevent stimulation and allow the pancreas gland to rest.

The current guidelines recommend the oral food intake should be tried as soon as possible, and beneficial effects or early enteral nutrition with mild AP have been reported in literature.

Then, early oral refeeding (EORF) after mild and moderate AP is beneficial, but the optimal timing and starting criteria are unclear. Even now, refeeding after mild and moderate AP is typically started until clinical symptoms have resolved and pancreatic enzymes are decreasing, in a successively increasing manner. The aim of this study is to evaluate length of hospital stay, clinical findings and complications for EORF with immediately full caloric intake in patients with mild and moderate AP.

DETAILED DESCRIPTION:
This is prospective, randomized, controlled, multicentre trial. Patients with mild and moderate acute pancreatitis (AP) will be randomly in two groups: group A: with early oral refeeding (EOR) with low fat solid diet (LFSD), started from the first day of admission in the hospital, and group B: with Nil Per Oral (NPO), until the symptoms, signs, inflammatory parameters of AP have resolved.

The primary and several secondary endpoints will be obtained and EORF with LFSD will improve the following measures of outcome:

1. Length of hospital admission (the primary endpoint)
2. Serum amylase, lipase, electrolytes, calcium, urea, creatinine, liver function tests, C-reactive protein (biomarker of inflammation), nutritional parameters (albumin, prealbumin, cholesterol, triglycerides) and full blood count - routine blood tests performed daily until normalization of serum lipase or until discharge.
3. Weight, at hospital admission and discharge, and at day 30 post-discharge clinic follow-up.
4. Systemic complications including hemodynamic instability, renal failure, intensive care admission, surgery, radiological and endoscopic procedures.
5. Pain and Analgesic requirement.
6. Local complications including pancreatic necrosis, abscess, pseudocyst.

ELIGIBILITY:
Inclusion Criteria:

* 1) Diagnosed of AP by at least two of these three criteria: compatible abdominal pain, amylase or lipase level superior in three-fold respective laboratory baseline levels, and suitable findings in imaging techniques (CT, ultrasound or MRI)
* 2) age > 18 years, sign consent form.

Exclusion Criteria:

* 1) pregnant o breastfeeding women;
* 2) abdominal pain lasting >96 horas before admission;
* 3) the possibility of poor oral intake for reasons other than AP;
* 4) Pancreatic neoplasm, endoscopic retrograde cholangiopancreatography or trauma etiology;
* 5) Chronic pancreatitis;
* 6) Randomization greater the 12 hours after admission

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | measured from onset of admission until time of actual discharge from hospital. Assessed between 1-10 days up to 14 days.
  Days

SECONDARY OUTCOMES:
Relapse of abdominal pain | measured from onset of admission until time of actual discharge from hospital. Assessed between 1-10 days up to 14 days, and during the follow up (1 month after discharge)
  Pain Scale: 0=No pain, 1=Very mild, 2=Discomforting, 3=Tolerable, 4=Distressing, 5=Distressing, 6=Intense pain, 7=Very intense pain, 8=Horrible pain, 9=Excruciating, 10=Unimaginable pain
Duration of fasting | 2-3 days approximately since the first day of hospital admission
  Days
Tolerance to food | 2-7 days approximately during hospital admission and during the follow up
  The patient's symptoms are controlled with the established treatment and the patient can eat at least 50% of the meals
Elevation of serum amylase or lipase | 2-4 days approximately during hospital admission after oral refeeding, until hospital discharge
  Elevation amylase or lipase level after oral refeeding
Intra-abdominal infection | 1 month
  Fever: temperature greater than 38 or positive cultures of blood or pancreatic necrosis
Death | During hospital stay (up to 1 day)
  Mortality
Operation rate | 2 month
  The rate of patients received operation for pancreatitis debridement

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ramírez-Maldonado, MD, Principal Investigator — Consorcio Sanitari del Garraf
Locations (1):
- Consorci Sanitari del Garraf, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The results of this trial will be published in an open access way and disseminates among medical societies
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From June 2019 the data will be available until publication
Access Criteria: Open accès publication

REFERENCES:
- [Background] Greenberg JA, Hsu J, Bawazeer M, Marshall J, Friedrich JO, Nathens A, Coburn N, May GR, Pearsall E, McLeod RS. Clinical practice guideline: management of acute pancreatitis. Can J Surg. 2016 Apr;59(2):128-40. doi: 10.1503/cjs.015015. PMID 27007094
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Bevan MG, Asrani VM, Bharmal S, Wu LM, Windsor JA, Petrov MS. Incidence and predictors of oral feeding intolerance in acute pancreatitis: A systematic review, meta-analysis, and meta-regression. Clin Nutr. 2017 Jun;36(3):722-729. doi: 10.1016/j.clnu.2016.06.006. Epub 2016 Jun 16. PMID 27346178
- [Result] Lodewijkx PJ, Besselink MG, Witteman BJ, Schepers NJ, Gooszen HG, van Santvoort HC, Bakker OJ; Dutch Pancreatitis Study Group. Nutrition in acute pancreatitis: a critical review. Expert Rev Gastroenterol Hepatol. 2016;10(5):571-80. doi: 10.1586/17474124.2016.1141048. Epub 2016 Mar 15. PMID 26823272
- [Result] Jacobson BC, Vander Vliet MB, Hughes MD, Maurer R, McManus K, Banks PA. A prospective, randomized trial of clear liquids versus low-fat solid diet as the initial meal in mild acute pancreatitis. Clin Gastroenterol Hepatol. 2007 Aug;5(8):946-51; quiz 886. doi: 10.1016/j.cgh.2007.04.012. Epub 2007 Jul 5. PMID 17613280
- [Result] Eckerwall GE, Tingstedt BB, Bergenzaun PE, Andersson RG. Immediate oral feeding in patients with mild acute pancreatitis is safe and may accelerate recovery--a randomized clinical study. Clin Nutr. 2007 Dec;26(6):758-63. doi: 10.1016/j.clnu.2007.04.007. Epub 2007 Aug 24. PMID 17719703
- [Result] Li J, Xue GJ, Liu YL, Javed MA, Zhao XL, Wan MH, Chen GY, Altaf K, Huang W, Tang WF. Early oral refeeding wisdom in patients with mild acute pancreatitis. Pancreas. 2013 Jan;42(1):88-91. doi: 10.1097/MPA.0b013e3182575fb5. PMID 22836861
- [Result] Olah A, Romics L Jr. Enteral nutrition in acute pancreatitis: a review of the current evidence. World J Gastroenterol. 2014 Nov 21;20(43):16123-31. doi: 10.3748/wjg.v20.i43.16123. PMID 25473164
- [Result] Petrov MS, van Santvoort HC, Besselink MG, Cirkel GA, Brink MA, Gooszen HG. Oral refeeding after onset of acute pancreatitis: a review of literature. Am J Gastroenterol. 2007 Sep;102(9):2079-84; quiz 2085. doi: 10.1111/j.1572-0241.2007.01357.x. Epub 2007 Jun 16. PMID 17573797
- [Result] Zhao XL, Zhu SF, Xue GJ, Li J, Liu YL, Wan MH, Huang W, Xia Q, Tang WF. Early oral refeeding based on hunger in moderate and severe acute pancreatitis: a prospective controlled, randomized clinical trial. Nutrition. 2015 Jan;31(1):171-5. doi: 10.1016/j.nut.2014.07.002. Epub 2014 Jul 30. PMID 25441594
- [Result] Petrov MS, Pylypchuk RD, Uchugina AF. A systematic review on the timing of artificial nutrition in acute pancreatitis. Br J Nutr. 2009 Mar;101(6):787-93. doi: 10.1017/S0007114508123443. Epub 2008 Nov 19. PMID 19017421
- [Result] Li X, Ma F, Jia K. Early enteral nutrition within 24 hours or between 24 and 72 hours for acute pancreatitis: evidence based on 12 RCTs. Med Sci Monit. 2014 Nov 17;20:2327-35. doi: 10.12659/MSM.892770. PMID 25399541
- [Result] Larino-Noia J, Lindkvist B, Iglesias-Garcia J, Seijo-Rios S, Iglesias-Canle J, Dominguez-Munoz JE. Early and/or immediately full caloric diet versus standard refeeding in mild acute pancreatitis: a randomized open-label trial. Pancreatology. 2014 May-Jun;14(3):167-73. doi: 10.1016/j.pan.2014.02.008. Epub 2014 Mar 14. PMID 24854611
- [Derived] Ramirez-Maldonado E, Lopez Gordo S, Pueyo EM, Sanchez-Garcia A, Mayol S, Gonzalez S, Elvira J, Memba R, Fondevila C, Jorba R. Immediate Oral Refeeding in Patients With Mild and Moderate Acute Pancreatitis: A Multicenter, Randomized Controlled Trial (PADI trial). Ann Surg. 2021 Aug 1;274(2):255-263. doi: 10.1097/SLA.0000000000004596. PMID 33196485

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03829085/Prot_SAP_ICF_000.pdf